CLINICAL TRIAL: NCT04805411
Title: A Randomized, Double Blind, Placebo-Controlled Phase IIb Study to Evaluate the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Patients With Moderate-to-Severe Atopic Dermatitis (AD)
Brief Title: Subcutaneously CM310/Placebo in Patients With Moderate-to-Severe Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310AD002
Record Dates: First submitted 2021-03-14; First posted 2021-03-18 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-11

CONDITIONS: Moderate-to-severe Atopic Dermatitis
Keywords: Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose arm (Experimental): 600mg for 1st dose, and then 300 mg for 2-8nd doses, every 2 weeks, SC
  Interventions: Biological: CM310
- low-dose arm (Experimental): 300mg for 1st dose, and then 150 mg for 2-8nd doses, every 2 weeks, SC
  Interventions: Biological: CM310
- placebo (Placebo Comparator): placebo for 1-8 doses, every 2 weeks, SC
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CM310 — IL-4Rα monoclonal antibody
  Arms: High-dose arm; low-dose arm
Biological: Placebo — Placebo
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled phase IIb study to evaluate the efficacy, safety, PK, PD and immunogenicity of CM310 in moderate-severe AD subjects. The study consists of 3 periods, a up-to-4-week Screening Period, a 16-week randomized Treatment Period and a 8-week Safety Follow-up Period.

DETAILED DESCRIPTION:
Subjects will be required to apply moisturizers after ICF signed and continue throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as AD for at least 12 months before Screening, with below requirements: 1)EASI score ≥16 at Screening and Baseline; 2) IGA score ≥3 (0-5 points scale) at Screening and Baseline; 3) ≥10% BSA of AD involvement at Screening and Baseline; 4) Pruritus NRS average score ≥3 at Baseline.
* Inadequate response to topical medications.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Concurrent disease/status which may potentially affect the efficacy/safety judgement.
* Organ dysfunction.
* pregnancy.
* Other.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
EASI-75 | at Week 16
  Proportion of subjects with EASI-75 (≥75 percent improvement from baseline)

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) 0/1 | at week 16
  Proportion of subjects with IGA 0 or 1 (on a 6-point scale, range from 0-5 point, higher scores mean a worse disease severity) and a reduction from baseline of ≥2 points.
reduction of IGA from baseline of ≥ 2 points | at week 16
  Proportion of subjects with IGA 0 or 1 (on a 6-point scale, range from 0-5 point, higher scores mean a worse disease severity) and a reduction from baseline of ≥2 points.
The Eczema Area and Severity Index (EASI)-90 | at week 16
  Proportion of subjects with EASI-90 (≥90 percent improvement from baseline)
The Eczema Area and Severity Index (EASI)-50 | at week 16
  Proportion of subjects with EASI-50 (≥50 percent improvement from baseline)
Improvement of Numerical Rating Scale (NRS) | at week 16
  Proportion of subjects with improvement (reduction) of pruritus NRS of ≥4 points from baseline. The range of NRS is from 0 (no itch)-10 (worst imaginable itch).
Body Surface Area (BSA) | Baseline to Week 24
  Change from baseline in percent of BSA
Dermatology Life Quality Index (DLQI) | Baseline to Week 24
  Change from baseline in DLQI
Safety parameters | Baseline to Week 24
  Incidence of AE, abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Pharmacokinetics parameters | Baseline to Week 24
  trough concentration and exposure of CM310
Pharmacodynamics | Baseline to Week 24
  Serum Thymus and activation regulated chemokine (TARC)
Pharmacodynamics | Baseline to Week 24
  Total IgE level
immunogenicity | Baseline to Week 24
  Detection of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Hospital, Chongqing, Chongqing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Second Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Second Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital of Dermatology, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Second Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No